CLINICAL TRIAL: NCT04206254
Title: GP96 Heat Shock Protein-Peptide Complex Vaccine in Treating Patients With Liver
Brief Title: GP96 Heat Shock Protein-Peptide Complex Vaccine in Treating Patients With Liver Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cure&Sure Biotech Co., LTD (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-CH-19
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — glucose-regulated proteins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- gp96 group (Experimental): Patients only receive autologous gp96 vaccination after surgery (do not accept other anti-tumor treatments)
  6 times of gp96 vaccination are administered via subcutaneous injection in 25μg doses within 8 weeks after surgery. gp96 is administered once a week.
  Interventions: Biological: gp96
- Control group (No Intervention): Patients do not accept any anti-tumor treatmentsafter surgery

INTERVENTIONS:
Biological: gp96 — heat shock protein gp96-peptide complex made from a person's tumor cells may help the body build an effective immune response to kill tumor cells.
  Arms: gp96 group

SUMMARY:
This trial is to further study the safety and effectiveness of autologous gp96 treatment of liver cancer on the basis of preliminary work

DETAILED DESCRIPTION:
RATIONALE: heat shock protein gp96-peptide complex made from a person's tumor cells may help the body build an effective immune response to kill tumor cells.

Overall Goals:

- to evaluate the safety and induction of anti-tumor immunity by administration of an immunogenic human tumor cell vaccine, and assess immune response in relation to clinical outcome.

Primary Aim:

- to further evaluate effectiveness of autologous gp96 treatment of liver cancer on the basis of preliminary work.

Secondary Aims:

to study the immune response to vaccination, to monitor clinical responses , to further the safety of vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand the informed consent document; must sign the informed consent;
2. Aged 18 to 75 years old , sex is not limited;
3. must have undergone radical resection;AJCC TNM II、III、IV.
4. Availability of at least 1g tumor sample;
5. Adequate bone marrow function including the absence of lymphopenia (ANC > 1,500/ mm3; Hemoglobin > 10g/dL ; platelet count >100,000/mm3), adequate liver function (serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], alanine amino transferase [ALT] <2.5 times institutional upper limit of normals [IULNs] ), and adequate renal function (BUN and creatinine <1.5 times IULNs)
6. Agree to Surgical indications of Heart & lung and without the coagulation system disease
7. Patients could not have received previous anti-cancer treat before 4 weeks of gp96 treatment；

Exclusion Criteria:

1. Inability to comply with study-related procedures
2. Unavailability of at least 6 doses of vaccine
3. Severe allergies
4. Unstable or severe intercurrent medical conditions
5. Current diagnosis of Human Immunodeficiency Virus and Patients with active uncontrolled infection.
6. patients with any systemic disease needed to be treated with immunosuppressant or Corticosteroids.
7. Female patients who are pregnant or breastfeeding
8. Steroidal drugs are currently being used systemically.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-19 (Estimated); Primary Completion 2022-08-05 (Estimated); Study Completion 2023-08-05 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | 2 year

SECONDARY OUTCOMES:
Disease free survival | 5 year
changes in antigen specific T cells | within 3 days before the first vaccination and within 10 days after the last vaccination
  tumor antigen specific T cells are determined by IFN-γ Enzyme-linked Tumor antigen specific T cells will be determined by IFN-γ Enzyme-linked immunosorbent spot using the autologous tumor cell lysis as the antigen
Number of participants with adverse events related to gp96 immunotherapy | up to 3 months after vaccine completion
  A complete blood count will be requested before the first vaccination, after the second vaccination and after the last vaccination to monitor the side effect of gp96 immunotherapy. And blood chemistries will also be requested at the same time point for the same reason.And other adverse events related to gp96 immunotherapy will be recorded according to the NCI-CTCAE 5.0 criteria.
Overall survival | 5 year